CLINICAL TRIAL: NCT02262117
Title: A Prospective, Randomized, Controlled, Two-arm Study to Evaluate the Interest of the Pre-conceptional Endometrial Immune Profiling to Increase Birth Rates Through a Care Personalization in Reproductive Medicine Before IVF
Brief Title: Evaluate the Interest of the Pre-conceptional Endometrial Immune Profiling to Increase Birth Rates
Acronym: PRECONCEPTIO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P130929
Record Dates: First submitted 2014-10-07; First posted 2014-10-10 (Estimated); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Reproductive Medicine
Keywords: IVF, immune endometrial profile, treatment personalization
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | US Export: No

ARMS (2):
- standard care (Placebo Comparator): No specific treatment (standard care)
  Interventions: Other: standard care
- specific treatment (Experimental): As a deregulation has been diagnosed by immune analysis, a personalization of the medical care for this IVF/ICSI attempt will be dispensed Personalization of treatment should follow a step-to step decision tree.
  Interventions: Drug: specific treatment

INTERVENTIONS:
Other: standard care — No specific medical care
  Arms: standard care
Drug: specific treatment — Regarding the immune endometrial profiling, medical care (personalization of treatment) should follow a step by step decision tree.
  Arms: specific treatment

SUMMARY:
A prospective, randomized, controlled, open two-arm study to evaluate the interest of the pre-conceptional endometrial immune profiling to increase birth rates.

DETAILED DESCRIPTION:
Birth rates following an embryo transfer with a mean of two embryos transferred stagnate around 23% per transfer (annual report of the Agency of Biomedicine). Some estimates that half of infertile patients treated are partially or totally concerned by problem of inadequate uterine receptivity.

The investigators' hypothesis is that a pre-conceptional immune endometrial evaluation may increase significantly birth rates since successful implantation results from both the matching of a competent embryo within a competent endometrium.

The identification of endometrial biomarkers documenting the immune uterine environment during the implantation window would be able to improve the efficacy of ART through a personalization of treatment accordingly to the ability of the patients to receive their embryos. All patients with all inclusion criteria and no exclusion criteria will be included. Only patients with a deregulation (immune analysis) will be randomized.

ELIGIBILITY:
Inclusion Criteria:

* Infertile patients will be included at the beginning of their medical care in reproduction once the indication to perform either an IVF with or without ICSI has been established. The indication for IVF will be: tubal infertility, endometriosis, ovarian dysovulation with failure of intra-uterine insemination, idiopathic infertility The indication for ICSI will be: male infertility (oligo-astheno-teratospermia), previous failure of oocytes fertilization in IVF
* Patients should be younger than 38 years old (Age < 38)

  * with a normal ovarian reserve (AMH>1.5ng/ml, FSH<10 IU/l on day-3, antral follicles count (AFC) over 6 on day-3 of the cycle by ultrasound)
  * The range of the IVF or ICSI attempt should be lower than 3 or equal at 2 (first or second IVF/ICSI). If a live birth occurred in the past by IVF/ICSI, the range of the new attempt is 1.
* With a signed informed and consent form
* With medical insurance

Exclusion Criteria:

* Azoospermia or cryptozoospermia (Patient's partner)
* IVF/ICSI attempt scheduled in another ART unit
* Contraindication to any experimental treatment (Cortancyl, Intralipids, Human Chorionic Gonadotropin)
* Maternal serology positive for hepatite C or B

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2015-10-30 (Actual); Primary Completion 2024-03-22 (Actual); Study Completion 2024-04 (Actual)

PRIMARY OUTCOMES:
Live birth rate (without congenital abnormality or malformation)/transfer following the first (fresh) embryo transfer after uterine immune analysis | up to 18 months
  Live birth rate/transfer

SECONDARY OUTCOMES:
Ongoing pregnancy rate/transfer following the first embryo transfer at 12 weeks of amenorrhea | 12 amenorrhea weeks
  Ongoing pregnancy rate/transfer following the first embryo transfer
Number of physiological pregnancies after personalization | up to 18 months
  Physiological pregnancies are defined by a normal growth of the fetus and a birth at term.
Pregnancy rate/transfer following the first embryo transfer | 8 amenorrhea weeks
  Pregnancy rate/transfer following the first embryo transfer
Number of embryo implanted/number of embryos replaced) | at 8, 12 and 40 amenorrhea weeks
  Implantation rate
Number of early miscarriage in the first trimester | 12 amenorrhea weeks
  Number of early miscarriage in the first trimester
Number of late miscarriage | between 13 and 24 amenorrhea weeks
  Number of late miscarriage
Term of birth (for babies without congenital anormality or malformation) | up to 18 months
  Term of birth
Weight at birth | up to 18 months
  A weight of birth below the 10 percentile according to the table of reference with distribution of birth weight in function of the term of birth in the overall population define the intrauterine growth retardation (for babies without congenital anormality or malformation)
Number of prematurity (A birth below 37 weeks of amenorrhea defines the premature birth and before 28 weeks of amenorrhea the severe preterm birth) (for babies without congenital anormality or malformation) | between 28 and 37 amenorrhea weeks
  Number of prematurity (A birth below 37 weeks of amenorrhea)
Number of pre-eclampsia (defined as the association of hypertension over 14/9 mm of hg with proteinuria occuring during the pregnancy- this pathology is related to insufiscient invasion during the first trimester) | up to 18 months
  Number of pre-eclampsia (defined as the association of hypertension over 14/9 mm of hg with proteinuria occuring during the pregnancy- this pathology is related to insufiscient invasion during the first trimester)
Number of pathologic pregnancy included stillbirth and congenital abnormality | up to 18 months
  Number of pathologic pregnancy included stillbirth and congenital abnormality
Investigate if immunologic events studying on endometrial level have an impact on blood level or are independent. | up to 15 months
  Quantification by flow cytometry of circulating NK cells (CD56 +/CD16 -), T regulatory T cells (FoxP3) with study of the repretory of circulating and uterine NK receptors (NPp46, Nkp30, NKp44).

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie LEDEE, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Saint-Louis - Laboratoire MatriceLAb Innove, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ledee N, Petitbarat M, Dray G, Chevrier L, Kazhalawi A, Rahmati M, Vicaut E, Diallo A, Cassuto NG, Ruoso L, Prat-Ellenberg L. Endometrial immune profiling and precision therapy increase live birth rate after embryo transfer: a randomised controlled trial. Front Immunol. 2025 Feb 24;16:1523871. doi: 10.3389/fimmu.2025.1523871. eCollection 2025. PMID 40066441